CLINICAL TRIAL: NCT06305338
Title: Predicting Post-operative Intraocular Lens Tilt Using Optical Coherence Tomography Measurements and Partial Least Squares Regression Modelling
Brief Title: Predicting Intraocular Lens Tilt Using OCT Measurements and Partial Least Squares Regression Modelling
Acronym: Tilt
Status: Completed | Type: Observational
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-009
Record Dates: First submitted 2023-03-09; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Intraocular Lens; Cataract
Keywords: Tilt
MeSH Terms: conditions — Cataract | interventions — Tomography, Optical Coherence; Biometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Optical Coherence Tomography — the study releated measurements will be performed: IOLMaster 700, Casia 2 and Pentacam HR.
  Other Names: biometry (IOL Master700); Casia2; Pentacam HR

SUMMARY:
During cataract surgery an artificial intraocular lens (IOL) is implanted in the eye to replace the lens and to correct the refraction for distance vision. Misalignment of IOLs can cause severe loss of visual quality. Different types of misalignment are known. Tilt, one type of IOL misalignment is thought to play a negative role for the optical performance in eyes with IOL designs, especially, if they have aspheric, toric, or multifocal optics.

Various methods to measure IOL misalignments have been described. Studies assessing the IOL position have used subjective grading methods at the slit lamp examination or a Scheimpflug camera to assess IOL decentration and tilt. The subjective grading at the slitlamp may display considerable variability between examiners. This method is more qualitative than quantitative and does not allow fine resolution when reporting IOL tilt. The fact that the patient has no standardized target to focus on makes the method even less reliable. Scanning methods such as Scheimpflug photos require a very well dilated pupil exceeding 6mm to assess the IOL position. Additionally, it can be difficult to identify the anatomical structures of the eye that need to be used as points of reference. Scheimpflug camera images have been used for assessing IOL tilt previously, but erroneous results, often due to corneal magnification, have diminished their widespread use. Another possibility to assess tilt is the use of Purkinje reflexes. The light reflections of Purkinje images at ocular surfaces to evaluate ocular alignment have recently been utilized. Since light is reflected at all interfaces of media with a difference in refractive index, these reflections, called Purkinje images, can be used to assess tilt and decentration of IOLs. Two different clinically applicable Purkinjemeter system provide the measurement of IOL decentration and tilt. The main problem with Purkinje meters is accessibility, as there are only a few prototypes available worldwide.

The most recently developed method for tilt quantification is the use of optical coherence tomography. This method has several advantages compared to the previous methods: OCT based devices are available in most clinics, the resolution of modern OCT devices is high, and the measurements are reproducible.

Aim of this study is to measure tilt with two modern OCT based devices and one Scheimpflug camera and to predict the post-operative tilt using partial least squares regression. This method was developed by Wold and introduced to ophthalmology previously.

DETAILED DESCRIPTION:
During cataract surgery an artificial intraocular lens (IOL) is implanted in the eye to replace the lens and to correct the refraction for distance vision. Misalignment of IOLs can cause severe loss of visual quality. Different types of misalignment are known. Tilt, one type of IOL misalignment is thought to play a negative role for the optical performance in eyes with IOL designs, especially, if they have aspheric, toric, or multifocal optics. For example, in the case of aspheric IOLs, it appears that even slight amount of tilt may result not only in the loss of the effect of reducing spherical aberrations but in more severe cases even a worsening of the optical quality compared to spherical IOLs. In the case of toric IOLs, tilt introduces higher order aberrations potentially mimicking astigmatism. In the case of multifocal IOLs, tilt increases higher order aberrations, which leads to decreased visual quality.

Various methods to measure IOL misalignments have been described. Studies assessing the IOL position have used subjective grading methods at the slit lamp examination or a Scheimpflug camera to assess IOL decentration and tilt. The subjective grading at the slitlamp may display considerable variability between examiners. This method is more qualitative than quantitative and does not allow fine resolution when reporting IOL tilt. The fact that the patient has no standardized target to focus on makes the method even less reliable. Scanning methods such as Scheimpflug photos require a very well dilated pupil exceeding 6mm to assess the IOL position. Additionally, it can be difficult to identify the anatomical structures of the eye that need to be used as points of reference. Scheimpflug camera images have been used for assessing IOL tilt previously, but erroneous results, often due to corneal magnification, have diminished their widespread use. Another possibility to assess tilt is the use of Purkinje reflexes. The light reflections of Purkinje images at ocular surfaces to evaluate ocular alignment have recently been utilized. Since light is reflected at all interfaces of media with a difference in refractive index, these reflections, called Purkinje images, can be used to assess tilt and decentration of IOLs. Two different clinically applicable Purkinjemeter system provide the measurement of IOL decentration and tilt. The main problem with Purkinje meters is accessibility, as there are only a few prototypes available worldwide.

The most recently developed method for tilt quantification is the use of optical coherence tomography. This method has several advantages compared to the previous methods: OCT based devices are available in most clinics, the resolution of modern OCT devices is high, and the measurements are reproducible.

Due to the fact that tilt has an influence on visual quality, the prediction of the post-operative tilt could improve IOL power calculation significantly, especially for toric IOLs. In the literature, the prediction of tilt was shown to be acceptable for the orientation of tilt, but not for the amount of tilt. Furthermore, there is disagreement concerning the fact, if the amount of tilt increases or decreases after cataract surgery.

Aim of this study is to measure tilt with two modern OCT based devices and one Scheimpflug camera and to predict the post-operative tilt using partial least squares regression. This method was developed by Wold and introduced to ophthalmology previously.

ELIGIBILITY:
Inclusion Criteria:

* Planned cataract surgery in one or both eyes
* Above 21 years of age

Exclusion Criteria:

* Combined surgery (cataract plus glaucoma/vitreoretinal/corneal surgery)
* Best corrected distance visual acuity below 0.05 Snellen
* Pathologies that could have an influence on the post-operative tilt, such as pseudoexfoliation syndrome or previous ophthalmic trauma, or other reasons for phakodonesis.
* Previous ophthalmic surgery that could have an influence on post-operative tilt, such as pars plana vitrectomy
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who undergo planned cataract surgeries above 21 years
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
post operative IOL tilt | 8 weeks post cataract surgery
  Predicting the post-operative tilt using PLS regression

SECONDARY OUTCOMES:
Comparison of tilt prediction | 8 weeks post cataract surgery
  Bilateral comparison of tilt prediction
comparion of three measurement methods | 8 weeks post cataract surgery
  Comparison between the three measurement methods concerning amount of tilt, orientation of tilt and tilt prediction
Comparison of tilt pre- versus post operative | pre operative at screening and 8 weeks post cataract operation
  Change of tilt from pre-operatively to post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Nino Hirnschall, MD, Principal Investigator — JKU Linz
Locations (1):
- Matthias Bolz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No